CLINICAL TRIAL: NCT00467285
Title: Effect of Thiazolidinediones on Skeletal Health
Brief Title: Effect of Diabetic Medications on Bone Metabolism
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: ENDB-019-06S
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Osteoporosis; Type 2 Diabetes Mellitus
Keywords: Bone Density; C-telopeptide; Dual-Energy X-Ray Absorptiometry; N-telopeptide; Osteocalcin; Osteoporosis; Thiazolidinediones; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Osteoporosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and serum samples collected for the study will be spin and stored at -70 degree C and assays run intermittently
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: 140 subjects with type 2 diabetes on pioglitazone.
- Group 2: 140 subjects with type 2 diabetes not on pioglitazone.

SUMMARY:
Subjects with diabetes and pre-diabetes are said to have increased bone loss when compared to the general population. Pioglitazone a thiazolidinedione, is a Food and Drug Administration (FDA) approved oral anti-diabetic agent for the treatment of type 2 diabetes. Though there are many benefits for using thiazolidinediones in the treatment of type 2 diabetes, there is data that indicates that rosiglitazone therapy results in a significant decrease in total body bone mineral density in mice. Whether it is true in humans is not clear. If the animal data can be extrapolated to humans, thiazolidinediones may pose a significant risk of adverse effects on bone. This study hypothesizes that treatment with the thiazolidinedione pioglitazone may result in significant reduction in bone mineral density. The aims of this are: 1. to evaluate the effect of pioglitazone on skeletal health; 2. to measure the bone mineral density (BMD) of the spine and hip, as well as bone turnover markers, at different times of persons taking thiazolidinediones and others not taking them; 3. to determine the change in BMD and bone turnover markers within different groups at different times; and 4. to compare these changes.

DETAILED DESCRIPTION:
The prevalence rate of diabetes among veterans is 16% in general and 27% at out medical center compared to 6.3% among United States population. Subjects with diabetes and prediabetes said to have increased bone loss compared to the general population. Pioglitazone, a thiazolidinedione, is a Food and Drug Administration (FDA) approved oral anti-diabetic agent for the treatment of type 2 diabetes. Most of the pleiotropic effects of teh thiazolidinediones are beneficial in atherosclerosis and cancer, in addition to improving insulin resistance. Data from studies in mice show that rosiglitazone and pioglitazone therapy results in a significant decrease in total body bone mineral density was observed. Whether it is true in humans is not clear. There are no prospective studies to date. Subjects with diabetes are already at an increased risk for femoral fractures. If the animal data can be can be extrapolated to humans, thiazolidinedione pioglitazone may result in significant risk of adverse skeletal effects. This study hypothesizes that treatment with the thiazolidinedione pioglitazone may result in a significant reduction in bone mineral density. The aims of the study include: 1. To prospectively evaluate the effect of pioglitazone on skeletal health, we will study 140 subjects with diabetes receiving pioglitazone as part of their diabetes management and compare them with 140 diabetic controls (matched for age, sex, body mass index (BMI), smoking and alcohol history), not treated with pioglitazone. 2. To measure the bone mineral density by DXA at AP spine and hip, as well as bone turnover markers-procollagen type 1C-terminal propeptide (P1CP), and procollagen type 1N-terminal propeptide (P1NP), bone specific alkaline phosphatase, osteocalcin, plasma C-telopeptide (CTx) and N-telopeptide (NTx) at baseline, six and 12 months of follow-up. 3. To determine the change in BMD and bone turnover markers within each group from baseline to follow-up at six and 12 months. 4. To compare the changes in the BMD and bone turnover markers between groups at baseline and follow-up at six and 12 months.

Subjects: Prospectively study 140 subjects with type 2 diabetes and on pioglitazone, age, and sex matched controls.

Sample Size: The sample size is based on the primary objective of comparing the levels bone turnover markers and bone mineral density changes in diabetes with or without avandia.

Number of visits: 140 subjects with diabetes and on pioglitazone and 140 subjects with diabetes not on pioglitazone

1. Subjects will be studies at three visits.
2. The procedures to be done include assessment of bone mineral density measurement by dual X-ray absorptiometry (DXA), measurement of bone turnover markers like serum osteocalcin and urinary N-telopeptide after the informed consent. About 15ml (one tablespoonful) of blood will be drawn at each visit for the study.
3. All the baseline measurements will be repeated at 6 months and at one year.
4. Statistical analysis of the data will be done to compare the changes in bone turnover markers and bone mineral density between the two groups.

Site of the study: Overton Brooks VAMC Diabetics clinic and Primary care clinics.

If our hypothesis is proven correct, subjects with diabetes requiring thiazolidinediones should have bone turnover markers and BMD measurement at baseline and have serial follow up. Identification of subjects at high risk will allow health care providers to initiate necessary protective measures to protect the bone to decrease the fracture risk.

Potential Impact on Veterans Health Care: Identification of subjects at high risk will allow health care providers to initiate necessary preventive measures to protect the bone and decrease the risk of fractures, or avoid the use of TZDs altogether in select patients. Since the prevalence of diabetes is very high among veterans, evaluation of a possible risk of skeletal health with the use of pioglitazone is highly relevant to VA health care.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-55 years
* Gender: men and women
* Ethnicity: all ethnic groups
* 140 subjects with diabetes and no pioglitazone (recently started i.e. less than 3 months as well as those who have just initiated pioglitazone treatment)
* 140 control subjects (subjects with diabetes and not on pioglitazone) will be included
* The control subjects will be chosen to match age, sex, ethnicity and comparable smoking and alcohol history
* To avoid confusion factor of vitamin D and calcium intake, all the subjects will be given vitamin D and calcium supplements (USDA recommended doses)

Exclusion Criteria:

* Patients who are unable or unwilling yo give informed consent
* Immobilized or bed bound subject
* Subjects wil known diseases associated with disordered bone metabolism such as chronic renal insufficiency, chronic steroid use, primary hyperparathyroidism, untreated subclinical or clinical hyperthyroidism and Paget's disease. To identify subjects with decreased Glomerular filtration rate (GFR) even if creatinine is normal will be excluded (at the proposed study site, routine bm includes calculated GFR from the chemistry lab)
* Patients on medications that will alter bone metabolism will be excluded. They are glucocorticoids, gonadal hormones (testosterone in men and estrogen in women).
* Subjects with known history of chronic pancreatitis, pancreatectomy or malabsorption syndromes to avoid confounding factors known to affect vitamin D metabolism and indirectly bone mineral metabolism.
* Female patients with perimenopause or menopause: history of hypogonadism (History of ovariectomy or postmenopausal women) to avoid bone turn over changes secondary to hypogonadism. Perimenopausal women identifies by screening FSH and LH and excluding women with elevated FSH be excluded to avoid perimenopausal effect on bone turnover (women over 35 will still have a screening gonadal hormonal evaluation).

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: subjects with type 2 diabetes and less than 55 years with or without pioglitazone as part of their therapy for diabetes
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhashini Yaturu, MD, Principal Investigator — Albany VA Medical Center Samuel S. Stratton, Albany, NY

REFERENCES:
- [Result] Yaturu S, Dier U, Cui H, Mousa SA. Aspirin resistance in young men with Type 2 diabetes. Journal of diabetes mellitus. 2014 Jan 1; 4(1):72-6.
- [Result] Yaturu S, Davis J, Shi R. Decreased bone mineral density in young male veterans on Pioglitazone*. Journal of diabetes mellitus. 2012 Jan 1; 2(1):35-9.
- See also: journal web site with link to the article — http://dx.doi.org/10.4236/jdm.2012.21006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Endo-Research clinic
Pre-assignment Details: Young male veterans with type 2 diabetes with creatinine less than 1.4, aged less than 55 years
Groups:
- Group 1: 32 subjects with type 2 diabetes on pioglitazone.
- Group 2: 64 subjects with type 2 diabetes not on pioglitazone, less than 55 years old.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 32 | 64
Completed | 28 | 60
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone: 32 subjects with type 2 diabetes on pioglitazone.
- No Pioglitazone: 64 subjects with type 2 diabetes not on pioglitazone, less than 55 years old.
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | No Pioglitazone | Total
Number analyzed (Participants) | 32 | 64 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 64 | 96
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (2) | 49 (2) | 49 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 64 | 96
Ctx [Mean (Standard Deviation); unit: pg/mL] | 29 (2) | 19 (3) | 22 (3)

OUTCOME MEASURES:

1. Primary Outcome: Changes in BMD at Femoral Neck
Description: % changes in BMD ( BMD at Lumbar spine, femoral neck and 0.33 radius) and bone turn over markers in subjects with diabetes on pioglitazone compared to those who are not on Pioglitazone
Time Frame: 6 months
Population: 28 subjects on pioglitazone and 64 subjects not on pioglitazone
Measure: Mean (Standard Deviation); unit: percentage of change in BMD
Groups:
- Piogliazone: 32 Subjects with type 2 diabetes on Pioglitazone
- No Pioglitazone: 64 subjects with type 2 diabetes not on pioglitazone
Arm/Group | Piogliazone | No Pioglitazone
Number analyzed (Participants) | 28 | 64
percentage of change in BMD | -3.2 (0.25) | 0.25 (0.24)
Statistical Analysis 1: Comparison: Piogliazone vs No Pioglitazone; comparison of changes in BMD at 6months compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: CTx
Description: % Change in bone turnover markers at 6 month follow up compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Baseline Characteristics: Group 1: Mean age of 49 with mean BMI 0f 33.6 ± 5; HbA1C of 7.54
- Baseline Characteristics: Group 2: Mean age of 49 with mean BMI 0f 35.2 ± 5; HbA1C of 7.45
Arm/Group | Baseline Characteristics: Group 1 | Baseline Characteristics: Group 2
Number analyzed (Participants) | 28 | 64
pg/mL | 4.9 (2.1) | 4.8 (1.28)

3. Secondary Outcome: Osteocalcin
Description: % change at 6 month follow up compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Piogliazone | No Pioglitazone
Number analyzed (Participants) | 28 | 64
% change | -20.49 (2.5) | -12.44 (2)

4. Primary Outcome: Changes in BMD Total Hip
Description: % change at 6 month follow up compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change in BMD
Arm/Group | Piogliazone | No Pioglitazone
Number analyzed (Participants) | 28 | 64
% change in BMD | -3.5 (0.24) | -0.2 (0.21)

5. Secondary Outcome: Changes in CTx at Follow up
Description: % change in the levels of CTx at 6 months follow up compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Piogliazone | No Pioglitazone
Number analyzed (Participants) | 28 | 64
% change | 29 (2) | 19 (3)

6. Primary Outcome: Changes in BMD AP Spine
Description: % change in BMD at 6 month follow up compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change in BMD
Arm/Group | Piogliazone | No Pioglitazone
Number analyzed (Participants) | 28 | 64
% change in BMD | -0.1 (0.04) | 0.89 (0.1)

7. Primary Outcome: Changes in BMD 0.33 Radius
Description: % change in BMD at 6 month follow up compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change in BMD
Arm/Group | Piogliazone | No Pioglitazone
Number analyzed (Participants) | 28 | 64
% change in BMD | -3.8 (0.22) | -0.21 (0.4)

ADVERSE EVENTS:
Time Frame: adverse events not collected
Groups:
- Pioglitazone: Subjects on pioglitazone
- No Pioglitazone: Subjects not on pioglitazone
Arm/Group | Pioglitazone | No Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes